CLINICAL TRIAL: NCT02303093
Title: Non-Interventional Study on the Tolerability and Efficacy of IVIG
Acronym: GAM 10-06
Status: Completed | Type: Observational
Sponsor: Octapharma (Industry)
Responsible Party: Sponsor
Other Study IDs: GAM 10-06
Record Dates: First submitted 2014-11-20; First posted 2014-11-27 (Estimated); Results first posted 2021-06-29 (Actual); Last update posted 2021-06-29 (Actual); Status verified 2021-06

CONDITIONS: Primary and Secondary Immunodeficiency and Other Conditions Requiring Regular Administration of Octagam 5% or 10% IVIG
MeSH Terms: interventions — Panzyga

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Octagam: Patient receiving Octagam 5% or 10% IVIG
  Interventions: Biological: Octagam IVIG 5% or 10%
- Panzyga: Patient receiving panzyga
  Interventions: Biological: Panzyga

INTERVENTIONS:
Biological: Octagam IVIG 5% or 10% — Octagam IVIG 5% or 10%
  Groups: Octagam
Biological: Panzyga — Panzyga
  Groups: Panzyga

SUMMARY:
Non-Interventional Study on the Tolerability and Efficacy of octagam® 10%

DETAILED DESCRIPTION:
A Non-Interventional Study on the Tolerability and Efficacy of Octagam 5% or 10% or panzyga. Patients with any indication (replacement and immonomodulation) as prescribed by the treating physician. Marketed Octagam 5% or 10% or panzyga will be used according to the investigator prescription; intravenous (iv) administration.The primary objective is to detect and evaluate adverse drug reactions (ADRs) occurring during or after the administration of Octagam or panzyga in any indication, age group or treatment regimen, where a causal relationship to the administration of Octagam or panzyga is suspected.

ELIGIBILITY:
Inclusion Criteria:

* Any patient who needs to be treated with a product of this class because of his/her medical condition and whom the treating physician decides to prescribe Octagam or panzyga regularly, may be included.

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Any patient who needs to be treated with a product of this class because of his/her medical condition and whom the treating physician decides to prescribe Octagam or panzyga regularly, may be included.
Sampling Method: Non-Probability Sample
Enrollment: 344 (Actual)
Dates: Start 2011-08-01 (Actual); Primary Completion 2020-06-05 (Actual); Study Completion 2020-06-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lidia Cosentino, Study Director — Octapharma
Locations (34):
- Austria (6):
  - Octapharma Research Site, Gmunden
  - Octapharma Research Site, Graz
  - Octapharma Research Site, Klagenfurt
  - Octapharma Research Site, Oberndorf
  - Octapharma Research Site, Salzburg
  - Octapharma Research Site, Vienna
- Canada (5):
  - St. Paul's Hospital, Vancouver, British Columbia
  - Health Sciences Centre, Winnipeg, Manitoba
  - Hamilton Health Sciences, Hamilton, Ontario
  - St. Michael's Hospital, Toronto, Ontario
  - Hospital for Sick Children, Toronto, Ontario
- France (16):
  - Octapharma Research Site, Argenteuil
  - Octapharma Research Site, Béziers
  - Octapharma Research Site, Bourges
  - Octapharma Research Location, Caen
  - Octapharma Research Site, Caen
  - Octapharma Research Site, La Rochelle
  - Octapharma Research Site, Marseille
  - Octapharma Research Location, Marseille
  - Octapharma Research Center, Marseille
  - Octapharma Research Site, Montauban
  - Octapharma Research Site, Nantes
  - Octapharma Research Site, Nevers
  - Octapharma Research Site, Pessac
  - Octapharma Research Site, Pierre-Bénite
  - Octapharma Research Site, Rennes
  - Octapharma Research Site, Toulouse
- Spain (3):
  - Octapharma Research Site, Barcelona
  - Octapharma Research Site, Madrid
  - Octapharma Research Location, Madrid
- United Kingdom (4):
  - Octapharma Research Site, Leeds
  - Octapharma Research Site, London
  - Octapharma Research Site, Plymouth
  - Octapharma Research Site, Stafford

RESULTS

PARTICIPANT FLOW:
Groups:
- All Patients: All patients
Period: Overall Study
Arm/Group | All Patients
Started | 344
Completed | 344
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | All Patients
Number analyzed (Participants) | 344
Age, Continuous [Median (Full Range); unit: years] | 59 [0 to 93]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 160
  Male | 184
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 138
  More than one race | 0
  Unknown or Not Reported | 199

OUTCOME MEASURES:

1. Primary Outcome: Adverse Drug Reactions
Description: Number of patients with adverse drug reactions
Time Frame: up to one year
Measure: Count of Participants; unit: Participants
Groups:
- Octagam 5%: Octagam 5%
- Octagam 10%: Octagam 10%
- Octagam 5% and Octagam 10%, While Under Octagam 5%: Octagam 5% and Octagam 10%, while under Octagam 5%
- Octagam 5% and Octagam 10%, While Under Octagam 10%: Octagam 5% and Octagam 10%, while under Octagam 10%
- Octagam 10% and Panzyga, While Under Octagam 10%: Octagam 10% and Panzyga, while under Octagam 10%
- Octagam 10% and Panzyga, While Under Panzyga: Octagam 10% and Panzyga, while under Panzyga
Arm/Group | Octagam 5% | Octagam 10% | Octagam 5% and Octagam 10%, While Under Octagam 5% | Octagam 5% and Octagam 10%, While Under Octagam 10% | Octagam 10% and Panzyga, While Under Octagam 10% | Octagam 10% and Panzyga, While Under Panzyga
Number analyzed (Participants) | 139 | 183 | 11 | 11 | 11 | 11
Participants | 17 | 37 | 0 | 1 | 9 | 9

2. Secondary Outcome: Infection Occurrence
Description: Pool of PID/SID Patients: Influence of IVIG/SCIG Treatment. Frequency, intensity, and duration of infectious episodes assessed. At the last available assessment, the influence of study IVIG on the frequency, intensity, and duration of the infections.
Time Frame: Up to one year
Population: Number of patients in the safety population with the respective diagnosis who attended the respective visit. Not all patients attended respective visit.
Measure: Count of Participants; unit: Participants
Groups:
- Octagam 5% and Octagam 10%: Panzyga
- Octagam 10% and Panzyga: Octagam 10% and Panzyga
Arm/Group | Octagam 5% | Octagam 10% | Octagam 5% and Octagam 10% | Octagam 10% and Panzyga
Number analyzed (Participants) | 60 | 121 | 2 | 0
Participants
  Frequency of infections: Beneficial | 20 | 61 | 2 | 0
  Frequency of infections: Unchanged | 7 | 31 | 0 | 0
  Frequency of infections: Unfavourable | 0 | 5 | 0 | 0
  Frequency of infections: Missing | 33 | 24 | 0 | 0
  Intensity of infections: Beneficial | 20 | 55 | 2 | 0
  Intensity of infections: Unchanged | 7 | 40 | 0 | 0
  Intensity of infections: Unfavourable | 0 | 2 | 0 | 0
  Intensity of infections: Missing | 33 | 24 | 0 | 0
  Duration of infections: Beneficial | 20 | 50 | 2 | 0
  Duration of infections: Unchanged | 7 | 43 | 0 | 0
  Duration of infections: Unfavourable | 0 | 4 | 0 | 0
  Duration of infections: Missing | 33 | 24 | 0 | 0

ADVERSE EVENTS:
Time Frame: Approximately 12 months, observational study
Arm/Group | Octagam 5% | Octagam 10% | Octagam 5% and Octagam 10%, While Under Octagam 5% | Octagam 5% and Octagam 10%, While Under Octagam 10% | Octagam 10% and Panzyga, While Under Octagam 10% | Octagam 10% and Panzyga, While Under Panzyga
All-Cause Mortality (participants affected / at risk) | 1/139 | 0/183 | 0/11 | 0/11 | 0/11 | 0/11
Serious Adverse Events (participants affected / at risk) | 3/139 | 1/183 | 0/11 | 0/11 | 1/11 | 0/11
Other Adverse Events (participants affected / at risk) | 13/139 | 37/183 | 0/11 | 1/11 | 9/11 | 9/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Octagam 5% (N=139) | Octagam 10% (N=183) | Octagam 5% and Octagam 10%, While Under Octagam 5% (N=11) | Octagam 5% and Octagam 10%, While Under Octagam 10% (N=11) | Octagam 10% and Panzyga, While Under Octagam 10% (N=11) | Octagam 10% and Panzyga, While Under Panzyga (N=11)
Cardiogenic shock (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0
Embolism (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0
Hepatic enzyme increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0
Thrombosis (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Klebsiella infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Fluid overload (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 1 | NA
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Octagam 5% (N=139) | Octagam 10% (N=183) | Octagam 5% and Octagam 10%, While Under Octagam 5% (N=11) | Octagam 5% and Octagam 10%, While Under Octagam 10% (N=11) | Octagam 10% and Panzyga, While Under Octagam 10% (N=11) | Octagam 10% and Panzyga, While Under Panzyga (N=11)
Fatigue (General disorders) | 0 | 7 | 0 | 0 | 4 | 4
Chills (General disorders) | 0 | 6 | 0 | 1 | 1 | 0
Chest discomfort (General disorders) | 2 | 3 | 0 | 0 | 1 | 2
Feeling hot (General disorders) | 0 | 5 | 0 | 0 | 1 | 0
Malaise (General disorders) | 0 | 4 | 0 | 0 | 0 | 0
Influenza like illness (General disorders) | 0 | 4 | 0 | 0 | 0 | 0
PYREXIA (General disorders) | 0 | 0 | 0 | 1 | 1 | 0
ASTHENIA (General disorders) | 0 | 0 | 0 | 0 | 2 | 0
FEELING COLD (General disorders) | 0 | 3 | 0 | 0 | 0 | 0
CHEST PAIN (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
FEELING OF BODY TEMPERATURE CHANGE (General disorders) | 0 | 0 | 0 | 1 | 0 | 0
HEADACHE (Nervous system disorders) | 3 | 20 | 0 | 0 | 8 | 8
DIZZINESS (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 1
PARAESTHESIA (Nervous system disorders) | 0 | 0 | 0 | 0 | 2 | 0
DISTURBANCE IN ATTENTION (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
LETHARGY (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
TREMOR (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
NAUSEA (Gastrointestinal disorders) | 2 | 12 | 0 | 0 | 1 | 1
DIARRHOEA (Gastrointestinal disorders) | 0 | 5 | 0 | 0 | 0 | 1
VOMITING (Gastrointestinal disorders) | 2 | 3 | 0 | 0 | 0 | 1
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 0 | 3 | 0 | 0 | 0 | 2
ABDOMINAL DISCOMFORT (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 1 | 1
DYSPEPSIA (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 0 | 0
ABDOMINAL PAIN (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
PARAESTHESIA ORAL (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
PRURITUS (Skin and subcutaneous tissue disorders) | 0 | 3 | 0 | 0 | 1 | 0
HYPERHIDROSIS (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0 | 1 | 0
URTICARIA (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 1 | 2
COLD SWEAT (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
ERYTHEMA (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0 | 0 | 0
RASH PRURITIC (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 0 | 0 | 0
RASH (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 1
RASH ERYTHEMATOUS (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
FLUSHING (Vascular disorders) | 0 | 0 | 0 | 0 | 2 | 2
HYPERTENSION (Vascular disorders) | 2 | 0 | 0 | 0 | 1 | 0
HOT FLUSH (Vascular disorders) | 0 | 2 | 0 | 0 | 0 | 1
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 0 | 3 | 0 | 0 | 0 | 1
BACK PAIN (Musculoskeletal and connective tissue disorders) | 0 | 3 | 0 | 0 | 0 | 0
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 0 | 0 | 0
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 0 | 0 | 0
MUSCULOSKELETAL DISCOMFORT (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
DYSPHONIA (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 1
LOWER RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 | 2 | 0 | 0 | 0 | 0
BLOOD GLUCOSE INCREASED (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
INSOMNIA (Psychiatric disorders) | 0 | 0 | 0 | 0 | 2 | 1
SLEEP DISORDER (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1
CYANOSIS (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0
HYPERSENSITIVITY (Immune system disorders) | 0 | 2 | 0 | 0 | 0 | 0
DECREASED APPETITE (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-06-27): https://cdn.clinicaltrials.gov/large-docs/93/NCT02303093/Prot_000.pdf
  • Statistical Analysis Plan (2020-04-14): https://cdn.clinicaltrials.gov/large-docs/93/NCT02303093/SAP_001.pdf